CLINICAL TRIAL: NCT00729989
Title: Efficacy and Safety of Gastric Suctioning During Neonatal Resuscitation- A Randomized Clinical Trial
Brief Title: Efficacy and Safety of Gastric Suctioning During Neonatal Resuscitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project not funded
Sponsor: Benjamin T. Stevens (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor-Investigator, Benjamin T. Stevens, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200804774
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Distress
Keywords: Meconium Aspiration; Respiratory Distress; Meconium Stained Amniotic Fluid
MeSH Terms: conditions — Dyspnea; Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental)
  Interventions: Procedure: Gastric suctioning

INTERVENTIONS:
Procedure: Gastric suctioning — The stomach will be suctioned shortly following birth with an orogastric tube
  Arms: 2

SUMMARY:
The stomach of the newborn baby is often emptied soon after birth to prevent breathing problems (respiratory distress). Babies born with meconium-stained amniotic fluid and those with increased secretions associated with birth by C-section are thought to be at particular risk of breathing problems during the first minutes of life. Emptying the stomach by sucking out all its contents (gastric suctioning) is alleged to lessen the risk of aspiration and improve respiratory distress. This study will evaluate the usefulness of gastric suctioning during neonatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Term infant with meconium stained amniotic fluid or born by C-section

Exclusion Criteria:

* Prematurity
* Congenital Abnormality

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Respiratory Distress | Birth

SECONDARY OUTCOMES:
Apgar scores | Birth
Successful feeding/weight gain | Birth
Hospital length of stay | Birth

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Children's Hospital, Iowa City, Iowa, United States